CLINICAL TRIAL: NCT04160104
Title: Pre-procedure Modle Predicts Bowel Preparation Quality Prior Colonoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Other Study IDs: KT20190827-2
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Bowel Preparation; Colonoscopy
Keywords: Bowel preparation; BBPS
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: This cohort was used to establish the bowel preparation score (BPS).
  Interventions: Other: Questionnaire
- Validation cohort: This cohort was used to verify the bowel preparation score (BPS).
  Interventions: Other: Questionnair

INTERVENTIONS:
Other: Questionnaire — Patients were asked to complete a questionnaire before colonoscopy. Bowel preparation was subsequently assessed by single endoscopist in each center using Boston bowel preparation quality score (BBPS). Both univariate and multivariate logistic regression models were used to identify high-risk factors associated with IBP and a predicting model with the bowel preparation score (BPS) was developed in the training cohort.
  Groups: Training cohort
Other: Questionnair — Patients were asked to complete a questionnaire before colonoscopy. The predicting modle established by the training cohort will be used to assessing the preparation of validation cohort. The result will compared with endoscopists assessment of preparation.
  Groups: Validation cohort

SUMMARY:
Bowel preparation is closely llined to the quality of colonoscopy, inadequate bowel preparation (IBP) could lead to higher miss rate of adenomas, patients' discomfort and higher health expense. For the patients with possible IBP before the examination, it may be better to cancel the colonoscopy and repeat bowel preparation through modified or enhanced strategies. Thus, it is important to set up a model to predict the quality of bowel preparation individually.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90 years old who undergoing colonoscopy

Exclusion Criteria:

* failed colonoscopy because of technical chanllenge or poor tolerance of patients
* history of colorectal surgery
* prior finding of severe colonic stricture or obstructing tumor
* dysphagia
* compromised swallowing reflex or mental status
* significant gastroparesis or gastric outlet obstruction or ileum
* known or suspected bowel obstruction or perforation
* pregnancy
* unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective study involving two tertiary-centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Boston bowel preparation quality scale | 1 hour
  A 10-point scale (0 is worst, 9 is best)

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, China